CLINICAL TRIAL: NCT02896777
Title: Triple-arm Trial of pH (Tri-pH) Effect on Live Birth After ICSI
Brief Title: Triple-arm pH Comparison
Acronym: Tri-pH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Collaborators: Egyptian IVF Center (Other); Banon IVF Center Assiut, Egypt (Other)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Lab Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: pH Study
Record Dates: First submitted 2016-08-31; First posted 2016-09-12 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: In Vitro Fertilisation Outcome
Keywords: pH; IVF; live birth rate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transfer embryos from 7.20±0.02 pH (Experimental): In this arm, the intervention is to culture the inseminated oocytes in vitro in a pH of 7.2±0.02 from day 0 to 5/6 post IVF/ICSI. Then according to the result of the randomization, women will receive their embryos that will be cultured in this pH on either Day 3 or Day 5/6 post IVF/ICSI.
  Interventions: Other: Transfer embryo from pH 7.20±0.02 on either Day 3 or day 5/6
- Transfer embryos from 7.3±0.02 pH (Experimental): In this arm, the intervention is to culture the inseminated oocytes in vitro in a pH of 7.3±0.02 from day 0 to 5/6 post IVF/ICSI. Then according to the result of the randomization, women will receive their embryos that will be cultured in this pH on either Day 3 or Day 5/6 post IVF/ICSI.
  Interventions: Other: Transfer embryo from pH 7.3±0.02 either Day 3 or day 5/6
- Transfer embryo from 7.4±0.02 (Experimental): In this arm, the intervention is to culture the inseminated oocytes in vitro in a pH of 7.4±0.02 from day 0 to 5/6 post IVF/ICSI. Then according to the result of the randomization, women will receive their embryos that will be cultured in this pH on either Day 3 or Day 5/6 post IVF/ICSI.
  Interventions: Other: Transfer embryo from pH of 7.4±0.02 on either Day 3 or day 5/6

INTERVENTIONS:
Other: Transfer embryo from pH 7.20±0.02 on either Day 3 or day 5/6 — Post IVF/ICSI and according to the result of the randomization process, women will receive embryo from their oocytes that will be cultured in pH of 7.20±0.02.
  Arms: Transfer embryos from 7.20±0.02 pH
Other: Transfer embryo from pH 7.3±0.02 either Day 3 or day 5/6 — Post IVF/ICSI and according to the result of the randomization process, women will receive embryo from their oocytes that will be cultured in pH of 7.3±0.02.
  Arms: Transfer embryos from 7.3±0.02 pH
Other: Transfer embryo from pH of 7.4±0.02 on either Day 3 or day 5/6 — Post IVF/ICSI and according to the result of the randomization process, women will receive embryo from their oocytes that will be cultured in pH of 7.4±0.02 from day 0 to 5/6
  Arms: Transfer embryo from 7.4±0.02

SUMMARY:
The culturing human embryo in vitro is a process of myriad contributing elements. From these factors is the pH of embryo culture media, which is crucial for embryo development. The investigators plan to examine three different pH values of the culture media on the live birth rate of in vitro cultured human embryos.

DETAILED DESCRIPTION:
In vitro fertilisation laboratory is the black box in which early human embryo development of infertile couple occurs. This laboratory holds many variables such as incubator type, air quality, brands of culture media, culture temperature and the pH of culture medium. Despite the importance of the culture medium pH, there is no single RCT has examined its effect on live birth rate post in vitro fertilisation. The investigators of this study believe that leaving this crucial element to the wishes of large companies and media designers is unwise. This RCT aims to provide a conclusive answer on pH effect on live birth rate of in vitro cultured human embryos.

ELIGIBILITY:
Inclusion Criteria:

1. Women age of ≥ 18 to ≤ 40
2. BMI of ≤ 35 (After approval of the DMC on 19 Feb 2021 and the IRB thereafter, BMI is changed from ≤31 to ≤35 based on clinician request. DMC).
3. Normal responder (≥ 10 antral follicle count (AFC) during basal ultrasound examination)
4. PCOS
5. Women who have ≥ 1 year of primary or secondary infertility
6. Tubal factor (unilateral, bilateral obstruction or salpingectomy)
7. Normal semen parameters
8. Male factor: oligoasthenozoospermia or obstructive azoospermia
9. Women who are undergoing their first IVF or ICSI cycle or second IVF Cycle with previous successful attempt
10. Women who will undergo only fresh embryo transfer
11. Women who have normal endometrial thickness (> 7 mm) and echo-pattern at the time of hCG trigger
12. Women who have normal transvaginal ultrasound during the follicular phase (defined as no intra cavity pathology; e.g. submucousal myomas, polyps or septa)

Exclusion Criteria:

1. Women who had unilateral oophorectomy
2. Women who had uterine pathology or abnormality
3. Women or their husbands who had abnormal karyotyping
4. Women with history of recurrent abortions or repeated implantation failures
5. Women who had uncontrolled diabetes
6. Women with diagnosed or undiagnosed liver or renal disease
7. Women who had a history of severe ovarian hyperstimulation
8. Women who had history of malignancy or borderline pathology
9. Women who will not meet the inclusion criteria
10. Women who will refuse to participate in the study
11. Women with endometriosis
12. Patient undergoing PGS or PGD
13. Severe male factor and non-obstructive azoospermia.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2273 (Actual)
Dates: Start 2020-06-13 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
live-birth rate | > 20 weeks of gestation
  delivery of one or more viable infants > 20 weeks of gestation

SECONDARY OUTCOMES:
Biochemical pregnancy rate | within 7 weeks of gestation
  registered positive hCG ≥14 days after egg collection
Clinical pregnancy rate | ≥ 7 weeks of gestation
  presence of a foetal sac with a foetal heart beat on ultrasound > 7 weeks of presence of a foetal sac with a foetal heart beat on ultrasound > 7 weeks of gestation
Ongoing pregnancy rate | within 24 weeks of pregnancy
  Continued pregnancy after 20 weeks of gestation
Miscarriage rate | within 42 weeks of pregnancy
  Loss of pregnancy before week 20 of gestation
Term Live birth rate | ≥ 37 weeks of gestation
  Delivery of one or more viable infants ≥ 37 weeks of gestation
Live-birth-implantation rate | within 42 weeks of gestation
  Number of viable neonates per number of embryos transferred
Cumulative live birth after one fresh and one frozen transfer | within one year from randomization
  Registered live birth from one fresh and one frozen cycles
Preterm Birth rate | <37 weeks of gestation
  Delivery of one or more viable infants <37 weeks of gestation
Very preterm birth rate | <32 weeks of gestation
  Delivery of one or more viable infants <32 weeks of gestation
Still birth | 42 weeks after ICSI
  delivery of nonviable babies > 20 weeks of gestation
Low birth weight babies | 24 hours after delivery
  Viable neonate < 2500 gm within 24 hours of delivery
Congenital malformation | within 42 weeks of gestation
  delivery of congenitally malformed babies
Fertilisation rate | Within 18 hours of inseminating the oocyte
  Presence of 2 pronuclei17±1 hr post insemination/ICSI
Cleavage rate | Within 72 hours of inseminating the oocytes
  registered divided embryo per fertilised oocyte
High quality embryo on day 3 | Within 72 hours of inseminating the oocytes
  embryo of 7 or more appropriate-size blastomeres with < 10 fragmentation by volume per Istanbul Consensus
Blastocyst formation rate on day 5/6 | Within 5-7 days of inseminating the oocytes
  Formed blastocyst of any grade on day 5 or 6 per fertilized oocyte
High-quality blastocyst rate on day 5 | 5 Days of inseminating the oocytes
  Blastocyst of ≥ 3.1.1.grading per Istanbul Consensus on day 5
Cryopreservation rate on day 5/6 | 5-7 Days of inseminating the oocytes
  Number of cryopreserved blastocyst on day 5 and 6 per fertilized oocyte
Embryo utilization rate | 5-7 days post ICSI
  Embryo Utilization rate (number of cryopreserved embryos added to the transferred embryos per fertilized oocytes
Top-quality embryo utilization rate | 5-7 days post ICSI
  number of cryopreserved embryos added to the transferred embryos per fertilized oocytes

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Fawzy, Principal Investigator — Ibnsina Hospital
Locations (6):
- Egypt (6):
  - Qena Fertility Center, Qina, Qena Governorate
  - Royal Centre, Al Mansurah
  - Banon Assiut, Asyut
  - Egyptian IVF-ET Center, Cairo
  - Amshaj, Sohag
  - IbnSina IVF Center, Sohag

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fawzy M, Emad M, Wilkinson J, Mansour R, Mahran A, Fetih A, Abdelrahman M, AbdelGhafar H. Triple-arm trial of pH (Tri-pH) effect on live birth after ICSI in Egyptian IVF facilities: protocol of a randomised controlled trial. BMJ Open. 2020 Feb 4;10(2):e034194. doi: 10.1136/bmjopen-2019-034194. PMID 32024790